CLINICAL TRIAL: NCT00102518
Title: A Multi-Center, Open-Label, Safety and Tolerability Study of Flexible-Dose Oral Aripiprazole (2 Mg-30 mg) in the Treatment of Adolescent Patients With Schizophrenia and Child and Adolescent Patients With Bipolar I Disorder, Manic or Mixed Episode With or Without Psychotic Features
Brief Title: Aripiprazole Open-Label, Safety and Tolerability Study
Acronym: APEX 241
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31-03-241
Record Dates: First submitted 2005-01-29; First posted 2005-01-31 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-07

CONDITIONS: Schizophrenia; Bipolar Disorder
Keywords: Open Label; Aripiprazole; Bipolar I Disorder, Manic or Mixed Episode
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Mania | interventions — Aripiprazole

ARMS (1):
- NCT00102063 and NCT00110461 Subjects (Experimental): All subjects had either completed or had withdrawn from the double-blind extension phase of study NCT00110461 (OPDC 31-03-240) and study NCT00102063 (OPDC 31-03-239).
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — 2 to 30 mg/day orally (2, 5, 10, 15, 20, 25, or 30 mg/day); tablets in strengths of 2, 5, 10, and 15 mg were used to achieve desired doses
  Other Names: OPC-14597

SUMMARY:
The purpose of this study is to test the long-term safety and tolerability of aripiprazole in adolescent patients with schizophrenia, and child and adolescent patients with bipolar I disorder, manic or mixed episode.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent patients with schizophrenia, or child and adolescent patients with bipolar I disorder, manic or mixed episode

Exclusion Criteria:

* Patients with a co-morbid serious, uncontrolled systemic illness
* Patients with a significant risk of committing suicide

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 325 (Actual)
Dates: Start 2004-09; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (50):
- United States (50):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Costa Mesa, California
  - Local Institution, Fresno, California
  - Local Institution, Orange, California
  - Local Institution, Riverside, California
  - Local Institution, Rosemead, California
  - Local Institution, Sacramento, California
  - Local Institution, Temecula, California
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Altamonte Springs, Florida
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Hialeah, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, Miami, Florida
  - Local Institution, Orange City, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Atlanta, Georgia
  - Local Institution, Honolulu, Hawaii
  - Local Institution, Chicago, Illinois
  - Local Institution, Kansas City, Kansas
  - Local Institution, Lexington, Kentucky
  - Local Institution, Louisville, Kentucky
  - Local Institution, Lake Charles, Louisiana
  - Local Institution, Metairie, Louisiana
  - Local Institution, New Orleans, Louisiana
  - Local Institution, Somerville, Massachusetts
  - Local Institution, Clinton, Michigan
  - Local Institution, Kansas City, Missouri
  - Local Institution, Saint Charles, Missouri
  - Local Institution, Elmsford, New York
  - Local Institution, New York, New York
  - Local Institution, Olean, New York
  - Local Institution, Rochester, New York
  - Local Institution, Chapel Hill, North Carolina
  - Local Institution, Cleveland, Ohio
  - Local Institution, Lyndhurst, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Bala-Cynwyd, Pennsylvania
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Memphis, Tennessee
  - Local Institution, Bellaire, Texas
  - Local Institution, DeSoto, Texas
  - Local Institution, Houston, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Salt Lake City, Utah
  - Local Institution, Kirkland, Washington
  - Local Institution, Seattle, Washington
  - Local Institution, Spokane, Washington
  - Local Institution, Wauwatosa, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 157 centers in Argentina, Bulgaria, Croatia, India, Jamaica, Mexico, Romania, Russia, Serbia, South Africa, South Korea, Ukraine, and the United States between September 2004 and February 2007. A total of 325 subjects were screened for enrollment and all 325 subjects were enrolled.
Pre-assignment Details: All participants had previously completed NCT00102063 (OPDC 31-03-239, adolescents with schizophrenia) or had withdrawn from the double-blind extension phase of NCT00110461 (OPDC 31-03-240, children and adolescents with bipolar 1 disorder), both clinical studies of aripiprazole.
Groups:
- NCT00102063 and NCT00110461 Subjects: All subjects had either completed or had withdrawn from the double-blind extension phase of study 31-03-240 and study 31-03-239.
Period: Overall Study
Arm/Group | NCT00102063 and NCT00110461 Subjects
Started | 325
Completed | 238
Not Completed | 87

BASELINE CHARACTERISTICS:
Arm/Group | NCT00102063 and NCT00110461 Subjects
Number analyzed (Participants) | 325
Age Continuous [Mean (Standard Deviation); unit: years] | 15.02 (1.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140
  Male | 185
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44
  Not Hispanic or Latino | 281
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 34
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 38
  White | 206
  More than one race | 45
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: cm] | 164.09 (11.22)
Weight [Mean (Standard Deviation); unit: kg] | 63.19 (17.86)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.25 (5.21)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Experiencing SAEs
Description: Percentage of Subjects Experiencing SAEs. The incidences of SAEs are summarized by system organ class in CT-8.5.1; by system organ class and MedDRA preferred term and by system organ class, MedDRA preferred term, and severity.
Time Frame: Baseline and Week 23
Population: All enrolled subjects.
Measure: Number; unit: percentage of participants
Arm/Group | NCT00102063 and NCT00110461 Subjects
Number analyzed (Participants) | 325
percentage of participants | 6.2

2. Secondary Outcome: Change in Change in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: Change from baseline to the last scheduled post-baseline evaluation in PANSS total score, using observed cases (assessments performed at baseline and weeks 4, 12, and 26).
  This scale consists of symptom constructs (7 positive, 7 negative, 16 general psychopathology), each to be rated on a 7-point scale of severity with 1 being absent to 7 being extreme. Minimum score is 30 which is best outcome; maximum score is 210 for worse outcome.
Time Frame: Baseline and Week 26
Measure: Mean (Standard Deviation); unit: points
Arm/Group | NCT00102063 and NCT00110461 Subjects
Number analyzed (Participants) | 234
points | -7.5 (17.89)

3. Secondary Outcome: Change in Young Mania Rating Scale (Y-MRS) Total Score
Description: Change from baseline to last scheduled post-baseline evaluation in YMRS total score, using observed cases (assessments performed at baseline and weeks 4, 12, and 26).
  The Y-MRS consists of 11 items assessing the core symptoms of mania. Each item has 5 grades of severity. Minimum score on the scale is 0 (absent or normal). Maximum score on the scale is 60 (worse outcome or more severe symptoms).
Time Frame: Baseline and Week 26
Measure: Mean (Standard Deviation); unit: points
Arm/Group | NCT00102063 and NCT00110461 Subjects
Number analyzed (Participants) | 82
points | -7.74 (11.73)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected as spontaneous reports at all scheduled visit. Serious AEs were monitored until the subject's health returned to baseline status or other parameters returned to normal or were otherwise explained.
Description: Spontaneously reported at each visit in response to query of "How have you felt since your last assessment?"
Arm/Group | NCT00102063 and NCT00110461 Subjects
Serious Adverse Events (participants affected / at risk) | 20/325
Other Adverse Events (participants affected / at risk) | 230/325
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NCT00102063 and NCT00110461 Subjects (N=325)
Bronchitis acute (Infections and infestations) | 1
Hepatitis A (Infections and infestations) | 1
Electrocution (Injury, poisoning and procedural complications) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
Acute psychosis (Psychiatric disorders) | 1
Aggression (Psychiatric disorders) | 3
Bipolar disorder (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 1
Hallucination, auditory (Psychiatric disorders) | 1
Homicidal ideation (Psychiatric disorders) | 1
Impulsive behavior (Psychiatric disorders) | 1
Intentional self injury (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 2
Schizophrenia (Psychiatric disorders) | 4
Suicidal ideation (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NCT00102063 and NCT00110461 Subjects (N=325)
Nausea (Gastrointestinal disorders) | 25
Vomiting (Gastrointestinal disorders) | 18
Nasopharyngitis (Infections and infestations) | 18
Weight increased (Investigations) | 25
Increased appetite (Metabolism and nutrition disorders) | 15
Akathisia (Nervous system disorders) | 27
Extrapyramidal disorder (Nervous system disorders) | 48
Headache (Nervous system disorders) | 31
Somnolence (Nervous system disorders) | 42
Tremor (Nervous system disorders) | 19
Insomnia (Psychiatric disorders) | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No